CLINICAL TRIAL: NCT04556890
Title: Multi-target Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment for Major Depressive Disorder (MDD) and Comorbid Pain
Brief Title: Pain and Major Depressive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Juliana Corlier, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-000530
Record Dates: First submitted 2020-08-31; First posted 2020-09-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder; Chronic Pain
Keywords: TMS; MDD; Chronic Pain
MeSH Terms: conditions — Depressive Disorder, Major; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study design includes two different stimulation protocols consisting each of 30 sessions:
  A) Active rTMS treatment for depression (1800 pulses of active intermittent theta burst (iTBS) administrated at 120% MT to the left DLPFC) and sham treatment for pain at M1; B) Active rTMS treatment for both, depression and pain (1800 pulses of iTBS to left DLPFC followed by 1500 pulses of 10 Hz to M1)
Who Masked: Participant, Outcomes Assessor
Masking Description: All stimulation procedures will be double-blinded, with clinicians, raters and patients blinded to the type of administered treatment using a designated sham coil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS/Active iTBS DFPLC/Sham Pain M1 (Experimental)
  Interventions: Device: Active rTMS/Active iTBS DFPLC/Sham Pain M1
- Active rTMS/Active iTBS (Experimental)
  Interventions: Device: Active rTMS/Active iTBS

INTERVENTIONS:
Device: Active rTMS/Active iTBS DFPLC/Sham Pain M1 — Active rTMS treatment for depression (600 pulses of active intermittent theta burst (iTBS) administrated at 120% MT to the left DLPFC) and sham treatment for pain at M1
  Arms: Active rTMS/Active iTBS DFPLC/Sham Pain M1
Device: Active rTMS/Active iTBS — Active rTMS treatment for both, depression and pain (600 pulses of iTBS to left DLPFC followed by 600 iTBS + 1500 pulses of 10 Hz to M1
  Arms: Active rTMS/Active iTBS

SUMMARY:
This study will examine the effects of brain stimulation on pain symptoms associated with Major depressive disorder. This study will enroll 54 Subjects. Study subjects will be asked to complete surveys about their mood and well-being, 2 blood draws, 2 MRIs, 3 electroencephalograms, and receive 30 treatments of blinded transcranial magnetic stimulation. There is no control group as all subjects will receive some form of active treatment. Subjects are required to participate in 30-33 study visits and volunteer 40 hours of their time. Compensation for this study is $150 for completing all study activities.

DETAILED DESCRIPTION:
The main objective of the proposed study is to evaluate the therapeutic effect of multi-site repetitive Transcranial Magnetic Stimulation (rTMS) on chronic pain and inflammatory responses in Major Depressive Disorder (MDD). MDD is the leading cause of disability worldwide. One reason for the extraordinarily high burden of depression is painful somatic symptoms: more than half of MDD patients complain of moderate to severe pain that is associated with interference in function and unemployment and which can lead to opioid use disorder. The neuro-immune interaction is increasingly understood as the underlying mechanism of this comorbidity. Sustained psychosocial stress can cause a lasting increase in systemic inflammation, which may be a key mediator of chronic pain and depression. Pro-inflammatory cytokines have been linked to the dysregulation of signaling in the mesocorticolimbic system and affect-related circuits present in both chronic pain and depression. Meta-analyses have identified higher CRP, IL6, and TNFa among depressed patients. Additionally, CRP was found to be increasingly higher with higher number failed treatment trials, suggesting that treatment resistant depression (TRD) patients who qualify for rTMS tend to have higher inflammation than those who respond to pharmacological antidepressant treatment [6]. Further, baseline levels of transcriptional control pathways (TCP) related to immune or sympathetic activation and glucocorticoid insensitivity mediate experimentally induced depressed mood. Even though the inflammatory reaction may originate in the periphery, downstream effects can result in neuroinflammation and changes in neural network function through several immune-to-brain signaling pathways. Previous research has shown that functional connectivity between DLPFC and anterior cingulate cortex (ACC) also mediates neuroinflammation levels in ACC, and which was linked to depressive scores in chronic pain patients [8]. rTMS to the left dorsolateral prefrontal cortex (DLPFC) is a non-invasive neuromodulation technique that has proven clinical efficacy for MDD and rTMS to primary motor cortex (M1) has been demonstrated to reduce chronic pain, including fibromyalgia, neuropathic pain, headache and regional pain].

Based on these findings, the investigators hypothesize that combined rTMS to depression and pain targets will reduce both depressive and pain symptoms and will also result in an effective reduction of systemic inflammation. The proposed research will examine the effects of 30 neuro-navigated sessions of active vs. sham rTMS using 2 conditions: A) active rTMS at DLPFC and sham at M1; B) active rTMS at DLPFC and M1. This design will help to dissociate the impact of an antidepressant response on pain reduction (condition A), or whether the combined treatment (condition B) will result in a synergetic effect. The investigators will focus on pain types related to inflammation including fibromyalgia (FM) and ME/CFS, whose symptomatic profiles are closely overlapping with those of MDD and may thus preferentially respond to rTMS.

The investigators will combine the analysis of circulating pro-inflammatory cytokines with transcriptomic analyses, which may be even more sensitive to short-term changes. Functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) data will be used to assess biomarkers and mechanisms of action (MOA) of successful rTMS treatment for pain. The conceptualization of pain treatment in MDD at the brain network and systemic levels makes this study a highly innovative approach to neuropsychiatric research.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects must be between 18-75 years of age
* Language: Participants must speak English fluently, as demonstrated by verbal skills sufficient to answer questions at a level that assures adequate understanding of the study
* All subjects must be right-handed
* Must have confirmed diagnosis of moderate Major Depressive Disorder (single or recurrent episode), minimum score of 17 on the 17-item Hamilton Rating Scale for Depression (HAM-D17). No minimal MDD duration necessary for study participation
* Failure to respond to a minimum of 2 trials of antidepressant medication
* Failure to respond from at least two different agent classes
* Accompanied by at least two evidence-based augmentation therapies (Benzodiazepines do not count)
* Must have a trial of psychotherapy known to be effective in the treatment of MDD of an adequate frequency and duration*
* Must have a confirmed FM or ME/CFS diagnoses and moderate pain complaints, minimum score of 15 on the McGill Pain Questionnaire.
* Pain chronicity for at least 3 months prior to study enrollment.
* Subjects are willing and able to adhere to the treatment schedule and required study visits.

Exclusion Criteria:

* Are mentally or legally incapacitated, unable to give informed consent.
* Are pregnant.
* Have an active suicidal intent or plan.
* Have had prior Transcranial Magnetic Stimulation treatment.
* Have an infection or poor skin condition over the scalp where the device will be positioned.
* Have increased risk of seizure because of family history, stroke, or currently use medications that lead to increased risk for seizure.
* Psychotic depression or other acute or chronic psychotic symptoms or disorders (such as schizophrenia, schizophreniform or schizoaffective disorder) in the current depressive episode.
* Neurological conditions that include epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, having a history of repetitive or severe head trauma, or with primary or secondary tumors in the central nervous system.
* Presence of an implanted metallic and magnetic-sensitive medical device present in the body scan, including but not limited to a cochlear implant, infusion pump, implanted cardioverter defibrillator, pacemaker, vagus nerve stimulator, aneurysm clip, metal prosthesis, or metal aneurysm clips or coils, staples, or stents. (Note: Dental amalgam fillings are not affected by the magnetic field and are acceptable for use with transcranial magnetic stimulation and MRI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in depression scores | Through study completion, an average of 6 weeks
  Inventory of Depressive symptoms- Self (IDS-SR) scores will be analyzed as the primary outcome measure. The IDS-SR is a 30-item scale that measures various symptoms of depression. Each item is scored between 0-4. Severity of depression is associated with a higher score with scores ranging from 0 to 84.
Percent change in pain score | Through study completion, an average of 6 weeks
  McGill Pain questionnaire (MPQ) will be analyzed as the secondary outcome. MPQ is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain and effectiveness of an intervention. Scoring ranges from 0 to 78. A higher score is associated with greater pain.

SECONDARY OUTCOMES:
Levels of inflammatory markers and transcription factors | Through study completion, average of 6 weeks
  Specimen will be processed and compared based on levels of pro-inflammatory cytokines and transcription factors (TF) related to immune activation, sympathetic activation and glucocorticoid insensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No